CLINICAL TRIAL: NCT00853983
Title: An Open-Label, Phase I Study to Assess Absorption, Metabolism and Excretion of a Single Oral Dose of [14C]AZD0530 in Healthy Male Volunteers
Brief Title: Phase I Study to Assess Absorption, Metabolism & Excretion of a Single Oral Dose [14C]AZD0530 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mary Stuart, MD, Medical Science Director, Emerging Product Team 1, Oncology, AstraZeneca Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D8180C00013
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Healthy
Keywords: Healthy Volunteers; ADME
MeSH Terms: interventions — saracatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: [14C] AZD0530 — Solution, Oral, once

SUMMARY:
The aim of this study is to show how the body absorbs, metabolises and excretes the drug [14C]AZD0530. As for all clinical trials, safety and tolerability of the drug will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Regular Daily Bowel movements
* Veins suitable for cannulation or repeated venepuncture

Exclusion Criteria:

* Presence of any clinically significant illness
* Abnormal vital signs
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-03; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To characterise the absorption, metabolism and excretion of a single oral dose of 400mg [14C]AZD0530 | Multiple PK, Urine and faeces samples taken between predose to 240 hours post dose

SECONDARY OUTCOMES:
To evaluate the safety profile by assessment of adverse events, physical examination, pulse, blood pressure, clinical chemistry, haematology, urinalysis & ECG | From time of consent to last visit

CONTACTS AND LOCATIONS:
Overall Officials: Raj Chetty, MD, Principal Investigator — AstraZeneca, Clinical Pharamcology Unit, Alderley Park; Mary Stuart, MD, Study Director — AstraZeneca, Parklands, Alderley Park
Locations (1):
- Research Site, Alderley Park, Cheshire, United Kingdom